CLINICAL TRIAL: NCT00620425
Title: A Single-Center, Open-label, Single-Arm Study to Evaluate the Effects of Repeat Doses of Subcutaneously Delivered Sumatriptan Via the Intraject System of Local Injection Site Signs in Healthy Adult Subjects.
Brief Title: A Study on the Effects of Repeat Doses of Intraject® Sumatriptan on Local Site Signs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZX001-0703
Record Dates: First submitted 2008-01-02; First posted 2008-02-21 (Estimated); Results first posted 2012-07-17 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: sumatriptan; Intraject; Local Site Reactions
MeSH Terms: interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sumatriptan — injection
  Other Names: SUMAVEL(R) DosePro(R)

SUMMARY:
Intraject is a needle-free, single use, disposable, subcutaneous delivery system pre-filled with 6 mg sumatriptan. Healthy Individuals will be enrolled for a series of 3 injections over 2 days. Assessment of Local Site Signs will be recorded for up to 5 days, as needed.

DETAILED DESCRIPTION:
This study will evaluate the extent, persistence, and any cumulative effects on skin tissue by assessing local injection site reactions (bleeding, swelling, erythema, bruising) following repeated administrations of needle-free Intraject sumatriptan to the same anatomic site.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of child-bearing potential must agree to use acceptable birth control
* Have abdominal or thigh injection sites that have sufficient subcutaneous tissue for needle-free injection
* Fluent in the spoken and written English language
* Provide written informed consent to participate in the study and be willing to comply with the study procedures
* Non-tobacco user for at least 12 months prior to screening (all types of tobacco, including cigars)

Exclusion Criteria:

* A history, symptoms, or signs of ischemic cardiac, cerebrovascular, or peripheral vascular syndromes including ischemic or vasospastic coronary artery disease
* Other significant underlying cardiovascular diseases including uncontrolled hypertension
* Hemiplegic or basilar migraine
* A history or diagnosis of severe hepatic or renal impairment
* A history of epilepsy or seizure or other serious neurologic condition
* A history of allergy, anaphylaxis, or hypersensitivity to sumatriptan or any of its components or similar drugs
* A history of scleroderma (systemic sclerosis) or any skin condition that may adversely affect the injection or absorption of subcutaneously administered medications
* Tattoos, birthmarks or other significant skin discoloration in the thigh or abdominal area that are large enough to restrict injection site selection and/or evaluation
* Pregnancy or breast-feeding
* Have participated in a clinical trial or receipt of an experimental therapy within 30 days prior to dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Chandler, MD, Principal Investigator — Covance

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Every participant received SUMAVEL DosePro at time 0, 1 and 25 hrs. Every participant was monitored for the incidence and persistence of bleeding, bruising, swelling and erythema.
Period: Overall Study
Arm/Group | All Participants
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: The Number of Injections With Local Site Reactions (Bleeding, Swelling, Bruising and Erythema).
Description: Each of the 18 participants were injected three times (for a total of 54 injections)with Sumavel DosePro, and followed over three days.
Time Frame: -15 min, immediately Post-dose, and 1, 4, 8, 24, 48 and 72 hrs post-dose
Measure: Number; unit: injections
Units Other Than Participants: Injections
Groups:
- All Participants at -15 Min Pre-dose: Every participant received SUMAVEL DosePro at time 0, 1 and 25 hrs. Every participant was monitored for the incidence and persistence of bleeding, bruising, swelling and erythema.
- All Participants Immediately Post-dose; 1 hr Post-dose; 4 hr Post-dose; 8 hr Post-dose; 24 hr Post-dose; 48 hr Post-dose: These are the reactions relative to each injection (total of 3 injections in 18 participants).
- 72 hr Post-dose: Only 3 subjects were required to return on Day 4. Day 4 assessments included a 72 hour assessment for the first and second injections and a 48 hour assessment for the third injection.
Arm/Group | All Participants at -15 Min Pre-dose | All Participants Immediately Post-dose | 1 hr Post-dose | 4 hr Post-dose | 8 hr Post-dose | 24 hr Post-dose | 48 hr Post-dose | 72 hr Post-dose
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18 | 18 | 18 | 3
Number analyzed (Injections) | 54 | 54 | 54 | 54 | 54 | 54 | 39 | 6
injections
  Injections with Bleeding present | 0 | 51 | 0 | 0 | 0 | 0 | 0 | 0
  Injections with Bruising present | 0 | 0 | 0 | 1 | 3 | 4 | 10 | 1
  Injections with Swelling present | 0 | 39 | 18 | 0 | 0 | 0 | 0 | 0
  Injections with Erythema present | 0 | 9 | 39 | 37 | 18 | 13 | 2 | 0

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 6/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=18)
Paresthesia (Nervous system disorders) | 6 (6)
Headache (Nervous system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No